CLINICAL TRIAL: NCT05528471
Title: Dietary Fructose as a Mediator to Altered Liver Energy Metabolism and Oxidative Stress in Youth With Non-alcoholic Fatty Liver Disease: HELP THEM FLY.
Brief Title: Fructose and Liver Diseases in Youth: Help Them FLY
Acronym: FLY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Health services (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00049795
Record Dates: First submitted 2020-09-15; First posted 2022-09-06 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: Non-alcoholic fatty liver disease; Fructose; Hepatic energetics; Hepatic fat fraction; Adolescents
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Intervention group (Experimental): Iso-caloric and low fructose /low HFCS diet (~5% of total energy intake (TEI); HFCS max: 10-15% of total fructose intake) (n=35)
  Interventions: Other: Dietary intervention
- Control group (No Intervention): Iso-caloric with higher fructose diet (~10% of TEI; HFCS max 20-30% of total fructose intake) (n=35)

INTERVENTIONS:
Other: Dietary intervention — To compare an iso-caloric, low fructose diet (~5% of total energy intake (TEI); HFCS max: 10-15% of total fructose intake) to an iso-caloric, higher fructose diet (~10% of TEI; HFCS max 20-30% of total fructose intake) in adolescents with NAFLD. The 10% higher fructose diet is part of standard of care and is NOT the intervention.
  Other Names: Fructose intervention
  Arms: Intervention group

SUMMARY:
Obesity has been increasing all over the world. This has lead to a significant increase of a liver disease in children called non-alcoholic fatty liver disease (NAFLD). NAFLD is a liver disease that ranges from excess fat being stored in the liver to an inflamed and fatty liver with fibrosis to cirrhosis. NAFLD is thought to be caused by changes in energy, fat and carbohydrate metabolism induced by diets high in in processed foods. Sugary (especially high fructose corn syrup or HFCS) and fatty foods in processed foods have been shown to produce more insulin resistance, a factor that is thought to cause a fatty liver. Currently the main treatment for NAFLD is weight loss. However, it unknown the best way to achieve this. The investigator has shown previously that adolescents with NAFLD eat a lot of fatty and sugary foods, and that when they decrease the amount of foods they eat that contain HFCS, experience some improvements in insulin resistance and liver dysfunction even when they don't lose weight. The plan is to compare and contrast how two different diets (high vs low HFCS containing diets) may affect how much fat gets deposited in the liver and whether or not a lower diet in HFCS can help decrease liver damage in adolescents with NAFLD.

DETAILED DESCRIPTION:
Study Rationale: Non-alcoholic fatty liver disease (NAFLD) is a chronic liver disease estimated to occur in 10-20% of obese children and adults. High fructose and saturated fat intakes are thought to be major dietary factors contributing to over nutrition, insulin resistance, cardio-metabolic risk (e.g dysplipidemia, hypertension) and disease pathogenesis in adults and children with NAFLD . Although weight loss is the goal of treatment, there are currently no evidence based clinical guidelines regarding the specific dietary treatment needed for NAFLD. The investigator has shown previously that children and adolescents with NAFLD have diets rich in both total fructose (>10% of total energy intake) and high fructose corn syrup (20-50% of total fructose intake. These levels of intake were associated with increasing indices of liver dysfunction, insulin resistance and inflammation. In a recent pilot study, the investigator has showed that children with NAFLD experienced significant reductions in systolic blood pressure, percentage body fat, plasma markers of liver dysfunction (ALT, AST), cardio-metabolic risk (HOMA-IR, AI-IR, TG, Apo-B100) and alterations in body fat distribution in response to six months of an iso-caloric/low fructose diet (~5% of total kcal). High levels of fructose in the diet have been independently associated with insulin resistance, visceral adiposity, hepatic and skeletal muscle intramyocellular fat (IMF) deposition, altered hepatic mitochondrial function and energy utilization (ATP depletion), increased rates of de novo lipogenesis, inflammation, and hepatic fibrosis in both animal models and adults with NAFLD. While adult studies in NAFLD have related the impact of high intakes of HFCS to altered liver energetics (ATP production) and increasing insulin resistance and IMF , this has not be studied in obese children and adolescents with NAFLD. In addition, no information is available regarding the impact of dietary fructose reductions on these processes in either obese children, adolescents or adults with NAFLD. The plan is to use validated, non-invasive and safe methodologies such as Magnetic Resonance Imaging (MRI) and Magnetic Resonance Stimulation (MRS) to compare and contrast the effects of varying fructose intakes (low vs high) in iso-caloric diets on liver mitochondrial energetic (ATP production), hepatic and skeletal muscle fat content and markers of cardio-metabolic risk, liver dysfunction, insulin resistance, inflammation and oxidative stress in adolescents with NAFLD.

Hypotheses

1. Obese adolescents with NAFLD treated with a low fructose /low HFCS diet over 12 weeks, in the absence of weight loss, will result in significant improvements in indices of hepatic ATP production and reduced liver/ skeletal muscle fat deposition when compared to the effects of a higher fructose/higher HFCS diet.
2. Obese adolescents with NAFLD treated with a low fructose /low HFCS diet over 12 weeks, in the absence of weight loss, will result in significant improvements in indices of visceral and subcutaneous adiposity, insulin resistance and markers of liver and cardio-metabolic dysfunction, inflammation and oxidative stress when compared to the effects of a higher fructose/higher HFCS diet.

ELIGIBILITY:
Inclusion Criteria:

* obese boys and girls aged 12-18 years (Tanner Stage: III-V) with clinically diagnosed NAFLD

Exclusion Criteria:

1. all patients with a history of a known primary liver disease associated with steatohepatitis (Wilson disease, various metabolic disorders, viral hepatitis) (7);
2. All patients with a known primary diagnosis of Type 2 Diabetes or those on insulin;
3. Patients on medications known to cause hepatic steatosis (e.g., methotrexate, corticosteroids, valproic acid, statins);
4. Patients with evidence of bridging fibrosis (8); and
5. Patients with a known significant history of smoking or alcohol consumption (6, 9) and
6. Any patient undergoing an active weight loss program and/or who has received bariatric surgery for the treatment of obesity
7. Any participant with a cardiac pacemaker or with metal pins as this is a contraindication for MRS/MRI testing
8. Any participant of child bearing potential who is known to be pregnant (as this is a contraindication to MRS/MRI) testing. All females of child bearing potential will be asked to undergo a routine pregnancy test (urine) prior to MRS/MRI testing. This will be conducted in the baseline study visit
9. Any child with significant developmental delay or a significant co-morbidity that precluded the ability to participate in study procedures

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2015-04-30 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in 31P spectra from abdominal MRI scans in response to dietary intervention. | Change from baseline to 3 months
  Changes in area under the curve (AUC) for 31P spectra obtained from abdominal Magnetic Resonance Scan between baseline and 3 months between individuals and between study arms. We will calculate the difference (baseline value-3 months value) for each individual to determine the change from baseline. This will be done in both groups.

SECONDARY OUTCOMES:
Change in hepatic intramyocellular surface area in response to dietary intervention. | Change from baseline to 3 months
  Hepatic intramyocellular surface area (cm3/ht2) as measured by abdominal 1H1-Spectra obtained from Magnetic Resonance scans between baseline and 3 months between individuals and between study arms.The calculation for each value will (baseline value - 3 month value) for each individual. Unit have been provided in the description.
Change in visceral adipose tissue (VAT cm3/ht2) and subcutaneous adipose tissue (SAT cm3/ht2) surface area in response to the dietary intervention | Change from baseline to 3 months
  Changes in visceral adipose tissue (VAT) and subcutaneous adipose tissue (SAT) as measured from abdominal 1H1-abdominal MRI scans content/distribution between baseline and 3 months between individuals and between study arms.The calculation for each value will (baseline value - 3 month value) for SAT (cm3/height 2) and VAT (cm3/height2). . Unit have been provided in the description.
Change in markers of liver dysfunction in response to the dietary intervention | Change from baseline to 3 months
  Serum AST (U/L), ALT (U/L), GGT (U/L) between baseline and 3 months between individuals and between study arms. The calculation for each value will (baseline value - 3 month value) for each individual blood work. Unit have been provided in the description.
Change in cardio-metabolic risk factors in response to the dietary intervention | Change from baseline to 3 months
  Serum triglycerides (mmol/L) total cholesterol, HDL-and LDL cholesterol (mmol/L)) between baseline and 3 months between individuals and between study arms. The calculation for each value will (baseline value - 3 month value) for each individual blood work. Unit have been provided in the description.
Change in measures of insulin resistance in response to the dietary intervention | Change from baseline to 3 months
  Changes in markers of insulin resistance (serum insulin mU/L, HOMA-IR) between baseline and 3 months between individuals and between study arms. HOMA-IR is calculated by the following equation. HOMA-IR=fasting glucose in mmol/l*fasting insulin in μU/ml/22.5. The calculation for each value will (baseline value - 3 month value) for each individual blood work. Unit have been provided in the description.

CONTACTS AND LOCATIONS:
Overall Officials: Diana R Mager, PhD RD, Principal Investigator — University of Alberta
Locations (1):
- Clinical Research Unit, University of Alberta, Edmonton, Alberta, Canada